CLINICAL TRIAL: NCT02350387
Title: Efficacy of Eccentric Resistance Training in Persons With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Principal Investigator, Michael Bade, Assistant Professor, Regis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-010
Record Dates: First submitted 2015-01-20; First posted 2015-01-29 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Short Duration Exercise (Experimental): Participants randomized to this group will perform 4 sets of 8-15 repetitions of eccentric exercise using the Eccentron set at 50-80% of the participant's one repetition maximum.
  Interventions: Procedure: High Intensity Short Duration Exercise
- Low Intensity Long Duration Exercise (Experimental): Participants randomized to this group will perform 5-20 minutes of continuous eccentric exercise using the Eccentron set at 50% of the participant's one repetition maximum.
  Interventions: Procedure: Low intensity Long Duration Exercise

INTERVENTIONS:
Procedure: High Intensity Short Duration Exercise — Participants randomized to this group will perform 4 sets of 8-15 repetitions of eccentric exercise using the Eccentron set at 50-80% of the participant's one repetition maximum.
  Arms: High Intensity Short Duration Exercise
Procedure: Low intensity Long Duration Exercise — Participants randomized to this group will perform 5-20 minutes of continuous eccentric exercise using the Eccentron set at 50% of the participant's one repetition maximum.
  Arms: Low Intensity Long Duration Exercise

SUMMARY:
The purpose of this study is to determine if there are differences in balance, strength, functional performance and self-reported outcomes for subjects with knee osteoarthritis who complete a low intensity, long duration eccentric training program compared to those who complete a high intensity, short duration eccentric training program. This study will be utilizing the Eccentron (manufactured by BTE Technologies) for the performance of all eccentric exercise.

DETAILED DESCRIPTION:
Arthritis is the leading cause of disability in the United States. Osteoarthritis (OA) is the most common type of arthritis and affects nearly 27 million Americans. Knee OA is the most common type of osteoarthritis and is estimated to affect 42.1% of women and 31.2% of men over the age of 60.

Osteoarthritis is most likely multi-factorial with several underlying causes. It is no longer considered "a degenerative joint disease" but rather a process that involves dynamic biomechanical, biochemical, and cellular processes. It not only involves degeneration of the articular cartilage, but also inflammation of the synovium, changes to the underlying subchondral bone, and the development of osteophytes. Currently, it appears that numerous systemic factors can lead to the initiation of OA through different causal pathways . These systemic causes can then be amplified by local factors such as trauma or increased loading caused by obesity.

Currently, there is no "cure" for OA and attempts to find a disease modifying drug have been unsuccessful. Thus, treatment currently focuses on mitigating factors that are known to affect the radiographic progression of the disease as well as lead to activity limitation and participation restriction.9,10 Decreases in lower extremity strength are a major cause of activity limitations given the vital role of strength in activities of daily living.

One method that is used to mitigate progressing factors is through the use of an exercise program. Many types of exercise have been used successfully in the literature including resistance training. Resistance training can take many different forms such as isometric, isotonic (concentric and/or eccentric) or isokinetic with various intensities. Presently, there is little evidence for the use of eccentric training interventions for patients with knee OA. This study aims to further examine this type of resistance training for the OA population. Therefore, the purpose of this study is to examine the effects of low intensity, long duration eccentric resistance training and high intensity, short duration eccentric resistance training in individuals with knee OA. Ideally, this study will allow us to determine the overall effects of eccentric resistance training as well as the potential differences of the two types of eccentric resistance training.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be included in the study if they are:

* at least 55 years old,
* cognitively able to understand directions,
* able to ambulate at least 50 feet without stopping,
* are currently experiencing knee pain and
* meet at least 3 out of 6 criteria of the European League Against Rheumatism (EULAR) criteria for knee osteoarthritis diagnosis.

Exclusion Criteria:

Individuals will be excluded from the study if they have:

* a diagnosed medical condition that would limit physical ability, including acute or active fractures, myocardial infarctions, stroke,
* a traumatic brain injury within the last 6 months, or
* joint replacement within the last 12 months. Individuals with chronic neurological disorders limiting motion or present with any known contraindication for balance training will also be excluded from the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Isometric quadriceps strength as measured by a hand held dynamometer | Change from baseline to 8 weeks
  The primary outcome for this study is the change in quadriceps strength from baseline to 8 weeks (end of intervention) in both experimental groups.

SECONDARY OUTCOMES:
Lower extremity muscle strength as measured by a hand held dynamometer | Change from baseline to 8 weeks
  Trunk flexion/extension, Hip Abduction/Extension, Knee Flexion/Extension, and Ankle Plantarflexion and Dorsiflexion will be assessed at baseline and 8 weeks by a hand held dynamometer.
Timed Up and Go Test | Change from baseline to 8 weeks
6-minute Walk Test | Change from baseline to 8 weeks
Five times sit to stand test | Change from baseline to 8 weeks
Balance (assessed utilizing the romberg, sharpened romberg, one-legged stance test, functional reach test, and step test) | Change from baseline to 8 weeks
  Balance will be assessed utilizing the romberg, sharpened romberg, one-legged stance test, functional reach test, and step test.
Arthritis Impact Measurement Scale (AIMS) | Change from baseline to 8 weeks
Pain and muscle soreness ( assessed utilizing a numeric pain rating scale) | At the beginning of every treatment session and following every treatment session for the 8 week intervention
  Pain and muscle soreness will be assessed utilizing a numeric pain rating scale at the beginning and end of every treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bade, PT, PhD, Principal Investigator — Regis University
Locations (1):
- Regis University, Denver, Colorado, United States